CLINICAL TRIAL: NCT05279521
Title: The Effect of Interventional Pulmonary Rehabilitation Exercise on the Psychological Distress, Self-efficacy, and Quality of Life of Patients With Advanced Lung Cancer.
Brief Title: The Effect of Interventional Pulmonary Rehabilitation Exercise With Advanced Lung Cancer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 202103103RIND
Record Dates: First submitted 2022-02-16; First posted 2022-03-15 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Lung Cancer; Pulmonary Rehabilitation; Exercise; Lung Adenocarcinoma; Lung Tumor; Lung Neoplasms; Advanced Lung Cancer; Self Efficacy; Quality of Life; Psychological Distress
MeSH Terms: conditions — Lung Neoplasms; Motor Activity; Adenocarcinoma of Lung | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Mandatory exercise the lung rehabilitation exercise is divided into three parts: upper and lower limb muscle strength, endurance training and breathing training skills. It lasts for eight weeks of exercise training, and the exercise frequency is: three times a week.
  Interventions: Behavioral: pulmonary rehabilitation exercise
- Control group (No Intervention): Voluntary exercise the lung rehabilitation exercise is divided into three parts: upper and lower limb muscle strength, endurance training and breathing training skills. It lasts for eight weeks of exercise training, and the exercise frequency is: three times a week.

INTERVENTIONS:
Behavioral: pulmonary rehabilitation exercise — The lung rehabilitation exercise is divided into three parts: upper and lower limb muscle strength, endurance training and breathing training skills. It lasts for eight weeks of exercise training, and the exercise frequency is: three times a week.
  Other Names: exercise
  Arms: Experimental group

SUMMARY:
This study concluded that lung rehabilitation exercise programs can improve the psychological distress, self-efficacy, quality of life, six-minute walk distance, muscle strength, and reduce the number of hospitalizations for patients with advanced lung cancer.

DETAILED DESCRIPTION:
Lung cancer is the top ten cause of cancer death in Taiwan. Since symptoms in the early stage are insidious, most patients are diagnosed in the advanced stage.

Chemotherapy and radiotherapy are often necessary because most of the advanced stage lung cancer has metastasized and multi-organ involved. The prolonged treatment course and side effects of the chemotherapy and radiotherapy, as long as the low survival rate, all impaired the quality of life. Recent studies have shown that exercise can improve the quality of life of cancer patients; therefore, the purpose of this study is to explore the effects of interventional lung rehabilitation exercises on psychological distress, self-efficacy and quality of life in patients with advanced lung cancer. The research is an interventional study. For the experimental group, lung rehabilitation exercise programs, including endurance training, muscle strength training and breathing training, were given; for the control group, a leaflet for lung rehabilitation exercise were provided. Random allocation software was used to randomly allocate cases to the experimental group and the control group. The patients were enrolled from the ward of the Department of Thoracic Medicine in a teaching hospital in north Taiwan. The estimated number of enrollment was 104. The structured questionnaire was used for data collection and analysis. The questionnaire contained 4 dimensions, including basic demographic characteristics, anxiety and depression scale, self-efficacy scale and quality of life scale. The data were collected at 4 time points; before the intervention (baseline measurement, T1), 4 weeks after the intervention (T2), 6 weeks after the intervention (T3), and 8 weeks after the intervention program (T4). At the same time, the six-minute walking distance and maximum strength training test of each case were measured at the baseline (T1) and 8 weeks after the intervention program (T4). We used the independent sample test,chi square test , Pearson correlation coefficient analysis and single-factor analysis of variance, and the generalized estimation equation for analysis of the psychological distress, self-efficacy, and quality of life between the two groups. This study concluded that lung rehabilitation exercise programs can improve the psychological distress, self-efficacy, quality of life, six-minute walk distance, muscle strength, and reduce the number of hospitalizations for patients with advanced lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years old, diagnosed with advanced lung cancer of stage III and IV lung cancer, and the Eastern Cooperative Oncology Group (ECOG) score of 0 and 1 points.
* Plans to receive treatment or has received treatment, including chemotherapy, targeted therapy, radiation therapy, or combination therapy.
* Those who agree to participate in the research and accept regular follow-up interviews and fill in the written consent form after explaining and explaining the research process and rights in detail.

Exclusion Criteria:

* Those who are unaware or have cognitive impairment who cannot accept the questionnaire interview.
* Unstable angina, arrhythmia, myocardial infarction diagnosis.
* History of epilepsy.
* Heart failure [New York Heart Association, NYHA class IV].

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2022-03-20 (Estimated); Primary Completion 2023-02-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
psychological distress | The data were collected at 4 time points; before the intervention (baseline measurement, T1), 4 weeks after the intervention (T2), 6 weeks after the intervention (T3), and 8 weeks after the intervention program (T4).
  Hospital Anxiety and Depression Scale , HADS .There are 14 items in this scale, including 7 items for anxiety and 7 items for depression. Each item has 4 options and is scored from 0 to 3. The higher the score, the higher the degree of anxiety or depression. Because the question does not contain physical symptoms, but emotional states, it is more likely to avoid false positives caused by cancer symptoms, so it is widely used in emotional evaluation and screening of cancer patients. A score higher than 9 in the anxiety section, or a score higher than 8 in the depression section, or a total score higher than 15 requires clinical attention.
self-efficacy | The data were collected at 4 time points; before the intervention (baseline measurement, T1), 4 weeks after the intervention (T2), 6 weeks after the intervention (T3), and 8 weeks after the intervention program (T4).
  General Self-Efficacy Scale,GSES.The GSES is a 10-item psychometric scale with scores for each item ranging from 1 (not completely correct) to 4 (including completely correct). Scores range from 10 to 40, with the highest score indicating higher self-efficacy.
quality of life Functional Assessment of Cancer Therapy-Lung | The data were collected at 4 time points; before the intervention (baseline measurement, T1), 4 weeks after the intervention (T2), 6 weeks after the intervention (T3), and 8 weeks after the intervention program (T4).
  Functional Assessment of Cancer Therapy-Lung,FACT-L.FACT-L, Version 4, is a combination of the 27-item FACT-General (FACT-G) and the 9-item Lung Cancer Subscale (LCS) Items include: physical health status, social/family health status, emotional stability status, Functional health status, additional concerns, lung cancer-related issues, the score ranges from 0 to 4, and the higher the final value, the higher the score on the scale, and the better the quality of life.

SECONDARY OUTCOMES:
6MWT | baseline (T1) and 8 weeks after the intervention program (T4).
  Six-minute Walking Test
maximum strength training test | baseline (T1) and 8 weeks after the intervention program (T4).
  maximum strength training test

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu WL, Chien JY, Lu YY, Liu KF. Nurse-supported hybrid home-based pulmonary rehabilitation improves psychological distress, quality of life, and functional performance in advanced lung cancer: A randomized controlled trial. Eur J Oncol Nurs. 2026 Feb 5;81:103130. doi: 10.1016/j.ejon.2026.103130. Online ahead of print. PMID 41666769